CLINICAL TRIAL: NCT07384403
Title: Evaluation of Linear and Volumetric Soft Tissue Changes Following the Application of Topical Oxygen Therapy Around Customized Healing Collars: Case Series
Brief Title: Application of Topical Oxygen Therapy Around Customized Healing Collar
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mulhem Ahmad, Principal Investigator Mulhem Ahmad, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: per3312026
Record Dates: First submitted 2026-01-25; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Soft Tissue; Healing Abutment Influence on Gingival Volume; Soft Tissue Healing; Dental Implant Healing
Keywords: Oxygen gel; volumetic change of soft tissue; implant
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Topical Oxygen therapy (Experimental): Participants will undergo a standardized preoperative assessment prior to second-stage implant surgery, including medical and dental history review, clinical and radiographic evaluation to confirm implant osseointegration, and oral hygiene assessment with reinforcement as needed.
  During the second-stage procedure, local anesthesia will be administered, followed by a crestal incision to access the implant site. After removal of the cover screw, a customized PEEK healing abutment will be placed.
  Immediately after abutment placement, Blue®M oral gel (Blue®M Europe BV, The Netherlands) will be applied around the healing collar and gently massaged into the peri-implant mucosa. Participants will continue topical application twice daily for 7 days.
  Standard postoperative care will be provided. Clinical evaluations will be performed at baseline, 7 days, and 21 days to assess soft tissue changes, patient-reported outcomes, and clinical photographs.
  Interventions: Procedure: topical oxygen therapy

INTERVENTIONS:
Procedure: topical oxygen therapy — Participants will undergo a standardized preoperative assessment prior to second-stage implant surgery, including medical and dental history review, clinical and radiographic evaluation to confirm implant osseointegration, and oral hygiene assessment with reinforcement as needed. During the second-stage procedure, local anesthesia will be administered, followed by a crestal incision to access the implant site. After removal of the cover screw, a customized PEEK healing abutment will be placed. Immediately after abutment placement, Blue®M oral gel (Blue®M Europe BV, The Netherlands) will be applied around the healing collar and gently massaged into the peri-implant mucosa. Participants will continue topical application twice daily for 7 days. Standard postoperative care will be provided. Clinical evaluations will be performed at baseline, 7 days, and 21 days to assess soft tissue changes, patient-reported outcomes, and clinical photographs.

SUMMARY:
The preservation and enhancement of peri-implant soft tissues are essential for the long-term success and esthetic integration of dental implants. Customized healing abutments have been introduced to support individualized soft tissue shaping; however, optimizing soft tissue healing around implants remains a clinical challenge. Oxygen plays a critical role in wound healing by promoting angiogenesis, fibroblast proliferation, and collagen synthesis. Topical oxygen therapy has shown promise in accelerating tissue regeneration, yet its application in oral implantology, particularly in conjunction with customized healing abutments, has not been adequately studied. This study aims to provide clinical evidence regarding the effectiveness of topical oxygen therapy in improving linear and volumetric soft tissue changes around dental implants. The findings may guide clinicians in refining soft tissue management protocols and contribute to establishing evidence-based practices in implant dentistry.

DETAILED DESCRIPTION:
Interventions

Preoperative Measures Prior to the second-stage surgical procedure, all participants will undergo a standardized preoperative assessment to ensure their suitability for implant exposure and subsequent healing abutment placement.

The following components will be systematically conducted:

1. Medical and Dental History Evaluation A comprehensive evaluation of each patient's medical and dental history will be performed to identify any systemic conditions or pharmacological agents that may compromise wound healing or elevate the risk of postoperative complications.
2. Clinical and Radiographic Assessment A detailed clinical examination will be undertaken to evaluate the thickness of the soft tissue, the width of keratinized mucosa, and the condition of the mucosa overlying the implant site. Radiographic assessment using periapical radiographs or cone-beam computed tomography (CBCT), where indicated, will be conducted to confirm successful osseointegration of the dental implant and to exclude any evidence of peri-implant pathology.
3. Oral Hygiene Evaluation and Instruction Oral hygiene status will be assessed using the Plaque Index. Patients will receive personalized oral hygiene instructions to ensure optimal plaque control before the surgical intervention. In cases where oral hygiene is deemed suboptimal, professional mechanical plaque removal (PMPR) will be provided, followed by re-evaluation prior to proceeding with the second-stage surgery.

Surgical Protocol

During the second-stage procedure, local anesthesia will be administered via infiltration using 2% lidocaine with 1:100,000 epinephrine. A mid-crestal or slightly palatal crestal incision will then be made to access the implant site.

Once osseointegration is clinically confirmed, the cover screw will be removed. Subsequently, a customized healing abutment(PEEK), appropriate to the implant diameter, will be placed and securely hand-tightened.

Application of Blue®M Gel:

Immediately following the placement of the healing abutment, Blue®M oral gel (Blue®M Europe BV, theNetherlands) will be applied circumferentially around the healing collar using a sterile microbrush. The gel will be gently massaged into the peri-implant mucosa and left in situ.

Postoperative instructions will include:

* Patients will be advised to refrain from rinsing or brushing the treated area for the first 12 hours.
* Blue®M gel application will be continued by the patient twice daily for 7 days postoperatively, in conjunction with standard oral hygiene measures.

Postoperative Instructions and Follow-Up Patients will receive standard postoperative instructions and will be prescribed 0.12% chlorhexidine mouthwash to be used twice daily for one week. Analgesics (e.g., ibuprofen 400 mg) will be administered as needed. If sutures are used, they will be removed after 7-10 days.

Patients will be clinically evaluated at baseline (day of second-stage surgery), day 7, and day 21 for the following:

Horizontal and linear Soft tissue change ,Patient-reported outcomes (pain, discomfort),Digital photographs .

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 21 years and above.

  * Indicated for customized healing collar placement after second-stage surgery.
  * Good general health.
  * Able and willing to provide written informed consent.
  * Committed to follow-up visits.

Exclusion Criteria:

* Individuals below 21 years old.
* Systemic diseases affecting healing.
* Smokers/tobacco users.
* Pregnant/lactating women.
* Medications affecting soft tissue healing.
* Chemotherapy/radiotherapy patients.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Soft tissue dimensional changes | baseline: preoperative and after 3 months and after 6 months
  Horizontal Tissue Linear Alterations were measured in millimeters by superimposing baseline and follow-up 3D digital models and calculating the Mean Buccal Change (MBC) and Mean Total Change (MTC) using software such as ImageJ, Geomagic, or MeshLab at standardized buccal reference points.
  Vertical Linear Tissue Alterations were quantified in millimeters by evaluating changes in Mesial Papillae Height Variation (mPHv), Distal Papillae Height Variation (dPHv), Papillae Height Variation (PHv), and Midfacial Height Variation (MFHv) through calibrated digital photography or intraoral scanning relative to fixed anatomical landmarks.
Pink Esthetic Score (PES) | baseline: preoperative and after 3 months and after 6 months
  determined by scoring seven soft tissue parameters (papillae, mucosal contour, level, color, and texture) from 0 to 2, based on clinical photographs compared with adjacent teeth, yielding a total score ranging from 0 to 14.

SECONDARY OUTCOMES:
Postoperative Pain | baseline: at day 1 , day 3 , day 10
  assesse using the Numerical Rating Scale (NRS), where patients rated their pain intensity from 0 (no pain) to 10 (worst imaginable pain), either verbally or through a visual analog form.
Wound Healing | Baseline : day 1 , day 3 ,day 10
  evaluated using the Modified Healing Index (MHI) as proposed by clinically scoring tissue color, swelling, exudate, necrosis, granulation, and epithelialization, with each parameter assigned a value and summed to reflect overall healing quality.

CONTACTS AND LOCATIONS:
Overall Officials: Mulhem ahmed, Principal Investigator — Cairo University; maie ismael, Study Chair — Cairo University; Mona Darhous, Study Director — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt